CLINICAL TRIAL: NCT01349946
Title: Diffusion Weighted Imaging Evaluation for Understanding Stroke Evolution Study-2 (DEFUSE-2)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Pittsburgh (Other); Northwestern University (Other); University of Utah (Other); Oregon Health and Science University (Other); St. Luke's Medical Center (Other); Queen's Medical Center (Other); Swedish Health Services (Unknown); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gregory W Albers, MD, Professor of Neurology, Stanford University
Other Study IDs: SU-02082011-7478; 10752; R01NS039325 (NIH)
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Diffusion and Perfusion Imaging Evaluation for Understanding Stroke Evolution Study 2 (DEFUSE 2) is a multi-center pilot study to determine if cerebral perfusion imaging can help identify which patients, who are ineligible for intravenous tissue plasminogen activator (iv tPA) therapy or have failed iv tPA therapy, are most likely to benefit from an endovascular clot removal procedure.

DETAILED DESCRIPTION:
Currently, the only approved therapy for acute stroke patients is a medication called tissue plasminogen activator (tPA). This medication is given as an intravenous infusion and can dissolve blood clots, thereby restoring blood flow to the brain. Early restoration of blood flow can prevent the permanent damage to the brain which typically occurs after a stroke. As a result, patients who achieve early restoration of blood flow have less disability than stroke patients in whom blood flow is not restored. Unfortunately, only a very small fraction of stroke patients is treated with tPA and benefits from tPA. Nationwide only 3 percent of stroke patients receive this therapy. The short treatment time-window is one of the main reasons that patients are not eligible for this treatment. Previously, tPA was only recommended in the 0 - 3 hour time window after stroke onset, but recent studies have shown efficacy our to 4 ½ hours. AHA guidelines now recommend treatment with iv tPA up to 4 ½ hrs. However, the number of stroke patients who will benefit from treatment remains small despite expansion of the time-window from 3 to 4 ½ hrs. This is the result of two main limitations of tPA. First, the majority of stroke patients present beyond the 4 ½ hour time-window and will therefore remain ineligible for treatment. Second, stroke patients who receive tPA do not always benefit because the treatment does not restore blood flow in all patients. Our research has shown that depending on the location of the blood clot, blood flow is restored in only 20 to 50% of stroke patients treated with tPA.

Patients with persistent blood vessel occlusions and no improvement in their clinical condition after receiving tPA or those arriving at the hospital outside the 4 1/2 hour time window routinely undergo mechanical clot removal to open an occluded blood vessel in the brain.

Mechanical clot removal increases the percentage of stroke patients who achieve recanalization, and as a result may increase the proportion of patients who have good clinical outcomes. However it is unclear for which stroke patients mechanical thrombectomy is most suitable. Although effective at removing blood-clots, it appears that mechanical clot retrieval is not beneficial for all patients. Whereas some patients benefit, others experience no effect, and yet others are likely harmed by mechanical clot retrieval. In order to avoid harm and maximize benefit it is important to know, prior to initiation of the mechanical clot retrieval procedure, if the procedure is likely to result in a clinical improvement. The investigators hypothesize that the response to mechanical clot retrieval can be predicted based on characteristics of an MRI scan obtained just prior to the retrieval procedure. The investigators hope to learn if new MRI techniques can help identify which patients are most likely to benefit from mechanical clot removal after receiving tPA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Clinical diagnosis of ischemic stroke and a score of 5 or more points in the NIHSS.
3. Planned to undergo intra-arterial (IA) therapy for acute hemispheric stroke (Either as primary therapy or as adjuvant therapy following intravenous tPA treatment)
4. Planned to have a standard MRI including perfusion imaging and MR angiography of the circle of Willis (MRA) prior to IA therapy
5. Intra-arterial thrombectomy can be started within 90 minutes of completion of MRI scan and within 12 hours of symptom onset. (Start of IA therapy is defined as the time of insertion of the femoral artery sheath; Time of brain scan is defined as the time that the scan is completed)
6. Able to obtain informed consent (informed consent should be obtained prior to the baseline MRI scan).

Exclusion Criteria:

1. Any pre-existing neurological illness resulting in a modified Rankin Scale Score of 3 or higher prior to the qualifying stroke
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population includes those people with acute ischemic stroke
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2008-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
NIHSS Score | 30 days

SECONDARY OUTCOMES:
Modifies Rankin Score | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory W Albers, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - Stanford University School of Medicine, Stanford, California
  - The Queen, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Swedish Hospital, Seattle, Washington

REFERENCES:
- [Result] Lansberg MG, Straka M, Kemp S, Mlynash M, Wechsler LR, Jovin TG, Wilder MJ, Lutsep HL, Czartoski TJ, Bernstein RA, Chang CW, Warach S, Fazekas F, Inoue M, Tipirneni A, Hamilton SA, Zaharchuk G, Marks MP, Bammer R, Albers GW; DEFUSE 2 study investigators. MRI profile and response to endovascular reperfusion after stroke (DEFUSE 2): a prospective cohort study. Lancet Neurol. 2012 Oct;11(10):860-7. doi: 10.1016/S1474-4422(12)70203-X. Epub 2012 Sep 4. PMID 22954705
- [Derived] Yu Y, Christensen S, Ouyang J, Scalzo F, Liebeskind DS, Lansberg MG, Albers GW, Zaharchuk G. Predicting Hypoperfusion Lesion and Target Mismatch in Stroke from Diffusion-weighted MRI Using Deep Learning. Radiology. 2023 Apr;307(1):e220882. doi: 10.1148/radiol.220882. Epub 2022 Dec 6. PMID 36472536
- [Derived] Marks MP, Lansberg MG, Mlynash M, Olivot JM, Straka M, Kemp S, McTaggart R, Inoue M, Zaharchuk G, Bammer R, Albers GW; Diffusion and Perfusion Imaging Evaluation for Understanding Stroke Evolution 2 Investigators. Effect of collateral blood flow on patients undergoing endovascular therapy for acute ischemic stroke. Stroke. 2014 Apr;45(4):1035-9. doi: 10.1161/STROKEAHA.113.004085. Epub 2014 Feb 25. PMID 24569816